CLINICAL TRIAL: NCT06681857
Title: Evaluation of Simultaneous Implant Placement and Maxillary Sinus Floor Elevation With Gelatin Sponge Versus Allogenic Demineralized Bone Matrix: (A Randomized Controlled Clinical Trial)
Brief Title: Maxillary Sinus Floor Elevation With Gelatin Sponge Versus Allogenic Demineralized Bone Matrix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed Nagi Alghandour, Lecturer, Beni-Suef University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 27
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Maxillary Sinus Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group: Gelatin Sponge (Active Comparator): The surgical intervention will be executed under local anesthesia. After the elevation of the full-thickness mucoperiosteal flap over the lateral wall of the maxillary sinus, a circular lateral window will be created by sinus low-speed bur grinding of the cortical ring to guard against the Shniederian membrane violation, followed by its separation along the sinus floor, lateral walls and the boundaries of the window to elaborate a smooth superior membrane elevation.
  The created spaces beneath the elevated Shniederian membrane will be filled up by an absorbable gelatin sponge for the test group patients followed by the coverage of the side window with collagen membrane, secured with bone tacks to guard against the graft fibroblastic invasion.
  Interventions: Procedure: Sinus lifting
- Control group: Allogenic Demineralized Bone Matrix (Active Comparator): The surgical intervention will be executed under local anesthesia. After the elevation of the full-thickness mucoperiosteal flap over the lateral wall of the maxillary sinus, a circular lateral window will be created by sinus low-speed bur grinding of the cortical ring to guard against the Shniederian membrane violation, followed by its separation along the sinus floor, lateral walls and the boundaries of the window to elaborate a smooth superior membrane elevation.
  The created spaces beneath the elevated Shniederian membrane will be filled up by allogenic (DBM) for the control group patients, followed by the coverage of the side window with collagen membrane, secured with bone tacks to guard against the graft fibroblastic invasion.
  Interventions: Procedure: Sinus lifting

INTERVENTIONS:
Procedure: Sinus lifting — The implant osteotomy will be initiated by pilot drill entries followed by sequential drills via the radiographic stent's sleeves to position the fixtures precisely into the pre-determined recipient sites. The Implant stability quotient (ISQ) will then be measured using an Osstell device after attaching intelligent implant pigs. Finally, the mucoperiosteal flaps will be sutured in place with 4-0 Prolene.

SUMMARY:
The post-extraction pneumatization of the maxillary sinus often compromises the ability of the maxillary molar to the optimal recipient of dental implants as a consequence of the quantitative reduction of the vertical bone height and the reduced bone quality of the region posterior maxillary segment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes, with an age range of (25 to 55 years) with unilateral or bilateral edentulous posterior maxillary molar region with \ vertical residual bone height of (four to six millimeters), a minimal horizontal bone width of six millimeters bone width, acceptable interarch space, and fair inter-jaw anteroposterior, horizontal and vertical relationships.
2. Proper general health and oral hygiene.

Exclusion Criteria:

1. The presence of sinusitis, local sinus pathosis, or a systemic disease that would affect the final treatment outcomes, bone remodeling process, or maxillary sinus health.
2. Those patients with a history of previous bone graft, sinus lift, or failed implant.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Vertical bone gain | 6 months
  baseline and final outcome for measuring both groups' radiographic vertical bone height gain as a primary outcome aided by the (Blue-sky software) identification of four reference points along each implant buccal, palatal, mesial, and distal surface
Stability | 6 months
  Aided by the Osstell device, the authors will record the (ISQ) readings at implant placement and upon its exposure for prosthetic rehabilitation after six months as a secondary outcome. The mean (ISQ) of the maxillary sinus lift procedure would employ the mean of parallel and perpendicular (ISQ) readings to each implant long axis where one implant is inserted and the mean of the two implant readings when two implants are placed.
  The numerical data concerning the primary and secondary outcomes will be recorded, scheduled, and submitted for statistical analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-suef university, Banī Suwayf, Egypt